CLINICAL TRIAL: NCT03984071
Title: The Predictive Value of Estimated Glomerular Filtration Rate (eGFR) for Adverse Cardiovascular Events in the Hospital in Patients With ST-segment Elevation
Brief Title: The Predictive Value of eGFR for Adverse Cardiovascular Events in Patients With STEMI
Status: Completed | Type: Observational
Sponsor: Dongying Zhang (Other)
Responsible Party: Sponsor-Investigator, Dongying Zhang, Professor, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Other Study IDs: 2019-06-11
Record Dates: First submitted 2019-06-11; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Estimated glomerular filtration rate(eGFR) is significantly reduced in patients with ST-segment elevation myocardial infarction (STEMI). The aim of this study is to research that the incidence of adverse cardiovascular events (MACE) in patients with ST-segment elevation myocardial infarction is significantly higher when the glomerular filtration rate below a certain value.

DETAILED DESCRIPTION:
The investigators retrospectively analyzed the clinical data of 1157 patients with ST-segment elevation myocardial infarction. In-hospital adverse cardiovascular events (MACE) was defined as: cardiac arrest, cardiac rupture, malignant arrhythmia, and cardiac death. All the patients were divided into 3 groups according to the patient's estimated glomerular filtration rate(eGFR) (eGFR≥90ml/min/1.73m2; 90ml/min/1.73m2>eGFR≥60ml/min/1.73m2; eGFR<60ml/min /1.73m2). COX regression analysis and K-M survival curves are used to calculate the correlation between eGFR and in-hospital MACE.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with STEMI 2.Patients from whom informed consent has been properly obtained in writing prior to start of the trial

Exclusion Criteria:

* 1.Patients with previous myocardial infarction, congenital heart disease 2.Patients with liver disease, and renal failure 3.Patients with immunologic disease, malignant tumors, pregnancy, infection caused by various pathogens, chronic inflammatory disease, trauma.

Ages: 24 Years to 93 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: STEMI Patients
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac events | The median time of 7 days
  Relationship between reduced eGFR and in-hospital MACE